CLINICAL TRIAL: NCT01894204
Title: Frequency and Risk Factors of the Lung High Blood Pressure Post-embolique in the Fall of a First Episode of Idiopathic Pulmonary Embolism. Study " PADIS HTP "
Brief Title: Determine the Frequency of a HTPPE in 5 Years (± on 1 Year) After a First Episode of Idiopathic Pulmonary Embolism.
Acronym: PADIS-HTP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The maximum of inclusions was reached
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RB 12.161 - PADIS HTP
Record Dates: First submitted 2013-06-28; First posted 2013-07-10 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-05

CONDITIONS: HTPPE; Idiopathic Pulmonary Embolism
Keywords: HTTPE; Idiopathic Pulmonary embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HTPPE (Other): No drug and no placebo were used in this study. For all the patients who participated at the study PADIS-EP, somme exams must be performed.
  Interventions: Other: HTPPE

INTERVENTIONS:
Other: HTPPE — No drug and no placebo were used in this study. Some exams must be performed (DLCO - evaluation of the dyspnoea and pulmonary scintigraphy), and in function of the result of the pulmonary scintigraphy, the medical care of the patient will be different : negative pulmonary scintigraphy, stop of the explorations and taken care usual of the patients; positive pulmonary scintigraphy,realisation of a cardiac echography to estimate the presence or not of a not very probable, possible or likely HTP. The indication of the right cardiac catheterization is then put on the combination of the results of the cardiac echography and the evaluation of the dyspnoea.

SUMMARY:
Forward-looking troop established(constituted) by the patients having been included in the study " PADIS EP ", PHRC on 2006 and 2009, randomized checked(controlled), double-blind, comparing an anticoagulating treatment(processing) extended by coumadine versus placebo during 18 months at patients having had a first episode of EP idiopathique treated(handled) initially 6 months by anti-vitamin K.

ELIGIBILITY:
Inclusion Criteria:

* Patients having ended the study PADIS EP after the visit of the end of study and having signed the consent HTP.

Exclusion Criteria:

* Refusal to grant in writing to participate in the study PADIS HTP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2013-06-27 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Frequency of a HTPPE | 24 months

SECONDARY OUTCOMES:
Mortality and cause | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Francis COUTURAUD, PU-PH, Principal Investigator — CHRU de Brest
Locations (8):
- France (8):
  - CHRU de Brest, Brest
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CH de Lannion, Lannion
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Pontchaillou - Hôpital Sud, Rennes
  - Hôpital Yves Le Foll, Saint-Brieuc
  - Hôpital de Bellevue - CHU de Saint-Etienne, Saint-Etienne
  - Hôpital Rangueuil, Toulouse

REFERENCES:
- [Derived] Fauche A, Presles E, Sanchez O, Jais X, Le Mao R, Robin P, Pernod G, Bertoletti L, Jego P, Parent F, Lemarie CA, Leven F, Le Roux PY, Salaun PY, Nonent M, Girard P, Lacut K, Savale L, Melac S, Guegan M, Mismetti P, Laporte S, Leroyer C, Montani D, Couturaud F, Tromeur C; PADIS-PE Investigators. Frequency and predictors for chronic thromboembolic pulmonary hypertension after a first unprovoked pulmonary embolism: Results from PADIS studies. J Thromb Haemost. 2022 Dec;20(12):2850-2861. doi: 10.1111/jth.15866. Epub 2022 Sep 25. PMID 36017744